CLINICAL TRIAL: NCT01246713
Title: Effect on Acetaminophen Metabolism by Liquid Formulations: Do Excipients in Liquid Formulation Prevent Production of Toxic Metabolites?
Brief Title: Effect on Acetaminophen Metabolism by Liquid Formulations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Harvard University (Other); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Michael Ganetsky, Assistant Professor of Emergency Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2010P000135; UL1RR025758 (NIH)
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Results first posted 2013-05-08 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-03

CONDITIONS: Acetaminophen Metabolism; Acetaminophen Poisoning; Drug Metabolism by Excipients
Keywords: acetaminophen; excipients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetaminophen solid formulation (Placebo Comparator): Subjects in this arm will receive a 15mg/kg dose of a solid acetaminophen formulation.
  Interventions: Drug: Acetaminophen solid formulation
- Acetaminophen liquid formulation (Active Comparator): Subjects in this arm will receive a 15mg/kg dose of a liquid acetaminophen formulation.
  Interventions: Drug: Acetaminophen liquid formulation

INTERVENTIONS:
Drug: Acetaminophen liquid formulation — Subjects in this arm will receive a 15mg/kg dose of a solid acetaminophen formulation.
  Arms: Acetaminophen liquid formulation
Drug: Acetaminophen solid formulation — Subjects in this arm will receive a 15mg/kg dose of a solid acetaminophen formulation.
  Arms: Acetaminophen solid formulation

SUMMARY:
The purpose of this study is to determine whether excipients in the liquid formulation of acetaminophen prevent the formation of the toxic metabolites of acetaminophen.

DETAILED DESCRIPTION:
Acetaminophen (APAP) poisoning is the most frequent cause of acute hepatic failure in the United States. Toxicity requires cytochrome P-450 bioactivation of APAP. Children are less susceptible to APAP toxicity; the current theory is that they have different metabolism than adults. However, children's liquid preparations of APAP contain excipients which have been shown to inhibit APAP bioactivation in vitro and in rodents. Children tend to ingest liquid preparations, which could potentially explain their decreased susceptibility instead of an intrinsically different metabolism. Further, our review of Poison Center epidemiologic data shows that liquid preparations are less toxic in adults. Our hypothesis is that excipients in liquid preparations inhibit the bioactivation of APAP. The design is a pharmacokinetic cross-over study in humans. Healthy adult subjects will be recruited for administration of therapeutic doses of APAP in capsule and liquid formulations. Plasma via a heplock will be collected at serial time points up to 8 hours and assayed for APAP and its metabolites. After a washout period, subjects will receive the same dose of APAP in the alternate preparation. The pattern of metabolites, indicating the activity of the bioactivating enzymes, will be compared. A significant difference in P-450 metabolites will support the hypothesis and provide preliminary data for studies in patients who have ingested potentially toxic doses of APAP. Ultimately, this work could support development of novel antidotal therapy for APAP overdose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer ages 18-40
* Not taking any chronic medications

Exclusion Criteria:

* Pregnancy
* Any history of liver disease
* Frequent alcohol use (2 or more drinks more than 4 times per week)
* Unable to provide informed consent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-12; Primary Completion 2011-05 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ganetsky, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Harvard - Thorndike Clinical Research Center at Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ganetsky M, Bohlke M, Pereira L, Williams D, LeDuc B, Guatam S, Salhanick SD. Effect of excipients on acetaminophen metabolism and its implications for prevention of liver injury. J Clin Pharmacol. 2013 Apr;53(4):413-20. doi: 10.1002/jcph.24. Epub 2013 Feb 22. PMID 23436315

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Whether subjects received the solid or liquid preparation initially was randomly chosen.
Groups:
- Solid Acetaminophen First, Then Liquid Acetaminophen: Study participants randomized to receive solid formulation first. They received a 15mg/kg dose of a solid acetaminophen formulation for pharmacokinetic sampling on first study day, then had at least a 2 week washout period, then received a 15mg/kg dose of a liquid acetaminophen formulation for pharmacokinetic sampling on subsequent study day.
- Liquid Acetaminophen First, Then Solid Acetaminophen: Study participants randomized to receive liquid formulation first. They received a 15mg/kg dose of a liquid acetaminophen formulation for pharmacokinetic sampling on first study day, then had at least a 2 week washout period, then received a 15mg/kg dose of a solid acetaminophen formulation for pharmacokinetic sampling on subsequent study day.
Period: First Acetaminophen Dosing (1 Day)
Arm/Group | Solid Acetaminophen First, Then Liquid Acetaminophen | Liquid Acetaminophen First, Then Solid Acetaminophen
Started | 6 | 9
Completed | 6 | 9
Not Completed | 0 | 0
Period: Washout (at Least 14 Days)
Arm/Group | Solid Acetaminophen First, Then Liquid Acetaminophen | Liquid Acetaminophen First, Then Solid Acetaminophen
Started | 6 | 9
Completed | 6 | 9
Not Completed | 0 | 0
Period: Second Acetaminophen Dosing (1 Day)
Arm/Group | Solid Acetaminophen First, Then Liquid Acetaminophen | Liquid Acetaminophen First, Then Solid Acetaminophen
Started | 6 | 9
Completed | 6 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants received a 15mg/kg dose of a solid acetaminophen formulation and a 15mg/kg dose of a liquid acetaminophen formulation separated by at least a 2 week washout period.
Arm/Group | All Study Participants
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Acetaminophen Metabolites
Description: Area-under-curve from time zero to 8 hours for APAP-cysteinate metabolite. Serum was collected just prior to and at hours 1, 2, 4, 6, and 8 after administration of the APAP dose.
Time Frame: 8 hours
Measure: Mean (Standard Error); unit: mcg.hr/ml
Groups:
- Acetaminophen Solid Formulation: Subjects in this arm will receive a 15mg/kg dose of a solid acetaminophen formulation. Results for APAP-cysteinate metabolite
- Acetaminophen Liquid Formulation: Subjects in this arm will receive a 15mg/kg dose of a liquid acetaminophen formulation. Results for APAP-cysteinate metabolite
Arm/Group | Acetaminophen Solid Formulation | Acetaminophen Liquid Formulation
Number analyzed (Participants) | 15 | 15
mcg.hr/ml | 2.411 (0.21) | 2.009 (0.17)

ADVERSE EVENTS:
Time Frame: Adverse even data was collected during the study period (first day of dosing, at least 2 week washout period, second day of dosing)
Groups:
- Solid Acetaminophen First, Then Liquid Acetaminophen: Participants in arm Solid Acetaminophen First: received a single 15mg/kg dose of a solid acetaminophen formulation first, and then a 15mg/kg dose of a liquid acetaminophen formulation after a 2 week washout period.
- Liquid Acetaminophen First, Then Solid Acetaminophen: Participants in arm Liquid Acetaminophen First: received a single 15mg/kg dose of a liquid acetaminophen formulation, and then a 15mg/kg dose of a solid acetaminophen formulation after a 2 week washout period.
Arm/Group | Solid Acetaminophen First, Then Liquid Acetaminophen | Liquid Acetaminophen First, Then Solid Acetaminophen
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/9
Other Adverse Events (participants affected / at risk) | 0/6 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No